CLINICAL TRIAL: NCT05015595
Title: Memantine for Refractory OCD Patients: a Pragmatic Double Blind, Randomized, Parallel Group, Placebo Controlled, Monocentric Trial
Brief Title: Memantine for Refractory OCD Patients
Acronym: MemaROCD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Massimo Pasquini, Associate Professor, PhD, MD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM11916B7477A1B6
Record Dates: First submitted 2021-07-13; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Refractory; Memantine; Augmentation medication
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memantine (Active Comparator): For thirty-two-week double-blind up-titration treatment period (from T0 to T4) each patient will receive a daily administration of Memantine up to 20mg/day.
  Subsequently, each patient will undergone to a double-blind down-titration treatment period for eight-weeks (from T4 to T5). At T4, the dose of Memantine will be reduced at 10mg/day due to safety reasons before the end of treatment (T5).
  Interventions: Drug: Memantine Oral Tablet
- Placebo (Placebo Comparator): For thirty-two-week double-blind up-titration treatment period (from T0 to T4) each patient will receive a daily administration of placebo 20 mg/day.
  Subsequently, each patient will undergone to a double-blind down-titration treatment period for eight-weeks (from T4 to T5). At T4, the dose of Placebo will be reduced at 10mg/day, following the study protocol, before the end of treatment (T5).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine Oral Tablet — Thirty-two-week double-blind up-titration treatment period (from T0 to T4): patients will be randomly assigned to one of two arms (Memantine or placebo) in a 1:1 ratio and will receive a daily administration of Memantine/placebo up to 20mg/day. Eight-week double-blind down-titration treatment period (from T4 to T5): At T4, the dose of Memantine/placebo will be reduced at 10mg/day due to safety reasons before the end of treatment (T5).
  Arms: Memantine
Drug: Placebo — Thirty-two-week double-blind up-titration treatment period (from T0 to T4): patients will be randomly assigned to one of two arms (Memantine or placebo) in a 1:1 ratio and will receive a daily administration of Memantine/placebo up to 20mg/day. Eight-week double-blind down-titration treatment period (from T4 to T5): At T4, the dose of Memantine/placebo will be reduced at 10mg/day due to safety reasons before the end of treatment (T5).
  Arms: Placebo

SUMMARY:
Obsessive-compulsive disorder (OCD) is a psychiatric syndrome characterized by unwanted and repetitive thoughts and repeated ritualistic compulsions aimed to decrease the distress. Symptoms can cause severe distress and functional impairment. OCD affects 2-3% of the population and is ranked within the ten leading neuropsychiatric causes of disability. Dysfunction of the cortico-striatal-thalamo-cortical circuitry (CSTC) has been implicated in OCD, including altered brain activation and connectivity. A complex dysregulation of glutamatergic signaling within the cortico-striatal circuitry has been proposed in OCD. Data obtained by several studies are suggesting of a reduced glutamatergic concentrations in the anterior cingulate cortex, combined with overactivity of glutamatergic signaling in the striatum and orbitofrontal cortex. A growing number of RCTs have assessed the utility of different glutamate-modulating drugs as an augmentation or monotherapy in OCD, including refractory patients. However, there are relevant variations in between studies in terms of treatment-resistance, comorbidity, age and gender of the patients. At the present time four RCTs are available on the efficacy of memantine as an augmentation medication for refractory OCD patients. Investigators intend to conduce a double-blind, randomized, parallel group, placebo-controlled, monocentric trial to assess the efficacy and safety of memantine, a low-to-moderate affinity noncompetitive NMDAR antagonist that is currently approved for the treatment of Alzheimer disease, as an augmentative agent to a SSRI in treatment of patients affected by severe refractory OCD. Study design consists of four distinct periods (52 weeks) including memantine titration, neuropsychological assessment and follow-up.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a severe and debilitating neuropsychiatric condition that has an estimated lifetime prevalence of 2.5-3.0% of the general population. Traditionally it is characterized by repetitive and intrusive thoughts (obsessions) and repeated ritualistic behaviours (compulsions) performed from affected individual to decrease the distress.

Conventionally OCD is driven by irrational beliefs (obsessions) considered as the product of a cognitive bias (including overestimation of threat, increased personal responsibility and thought-action fusion) and compulsions are rational avoidance response triggered by these irrational beliefs, a coping mechanism which neutralize anxiety and reduce the likelihood that fears will be realized. Recent data suggest that OCD is driven by a disruption in the balance between habit learning system and goal directed system. The habit learning system operates purely on the basis of historical information, whether or not actions were rewarded in the past, it can lead to behavioural inflexibility and in isolation is not an optimal way to make choices when faced with rapid changes in the environment; while goal directed system exerts control over habits in light of new information, including changes in the desirability of outcomes and changes to the contingency between actions and outcomes. Habits depend on recurrent circuits that connect cerebral cortex to the basal ganglia, termed cortico-striatal-thalamo-cortical circuitry (CSTC) loops. In the CSTC model of OCD, these loops become hyperactive or hyperconnected, self-exciting in a runaway positive feedback loop. This leads to the urge to perform compulsions, which in turn consolidates/strengthens the habit of performing compulsions, increasing the urge. Glutamate is the primary neurotransmitter within the implicated in OCD CSTC. Glutamatergic neurotransmission has a fundamental role for neuronal plasticity, learning, and memory. Excessive glutamate levels could lead to glutamate receptor hyperactivity or even excitotoxicity in neurons. However, in pathological conditions glutamate can act as a neuronal excitotoxin, leading to rapid or delayed neurotoxicity. Dysregulation of glutamatergic signaling within the CSTC has been proposed in OCD, with reduced glutamatergic concentrations in the anterior cingulate cortex, combined with overactivity of glutamatergic signaling in the striatum and orbitofrontal cortex. Increased glutamate levels have been measured in cerebrospinal fluid of OCD patients compared to healthy controls. Traditionally medications for OCD have targeted on serotonergic pathways. Serotonin reuptake inhibitors (SRIs); unfortunately, around 40% of patients with OCD do not achieve remission of their symptoms with SRIs. Even when switching to another selective serotonin re-uptake inhibitor or clomipramine, or when an atypical antipsychotic is added, the portion of refractory patients still remains around 30%. Refractoriness is defined by the fail of almost three trials with different Selective Serotonin Reuptake Inhibitors (SSRIs) at high dosages. In light of a possible role of glutamatergic signalling dysregulation in the OCD it is possible found candidates for augmentation strategy of OCD's therapy in glutamatergic drugs. This background has motivated interest in studying glutamate modulators in patients who are unresponsive to standard pharmacotherapeutic approaches. In particular, some studies using memantine and riluzole have been reported promising suggestions of benefit. Other studies have explored the role of stimulants and nutritional supplements such as inositol and N-acetylcysteine. Several clinical studies were conducted to evaluate the effect of glutamate-modulating drugs in OCD, however they significant differ in terms of treatment-resistance, comorbidity, age and gender of the patients. A recent review on the argument conduced by Marinova et al concluded that memantine is the compound most consistently showing a positive effect as an augmentation therapy in OCD. Moreover randomized placebo-controlled trials in clinical samples are necessary in order to draw definitive conclusions on the utility of glutamate-modulating drugs in OCD. Identifying and confirming the efficacy and safety of new therapeutic approaches for the OCD could be very useful also for improving disability and quality of life in these patients.

At the present time four RCTs are available on the efficacy of memantine as an augmentation medication for refractory OCD patients.

The main aim of this study is to conduce a double-blind, randomized, parallel group, placebo-controlled, monocentric trial to assess the efficacy and safety of memantine, a low-to-moderate affinity noncompetitive NMDAR antagonist that is currently approved for the treatment of Alzheimer disease, as an augmentative agent to a SSRI in treatment of patients affected by severe refractory OCD.

The second aim of the study is to evaluate the minimum effective dose of memantine in this patients and effects after drug withdrawal through follow up. The third aim is to investigated the effect of memantine on patients without cognitive impairment an improvement of cognitive functions.

Methods: A double-blind, randomized, parallel group, placebo-controlled, monocentric trial will be conduce over 52 weeks at the outpatient clinic of the Department of Human Neurosciences (Policlinico Umberto I, Rome). The study will be conducted in agreement with the Declaration of Helsinki and its subsequent revisions. At the same time the study will be subject to the ethics committee of Policlinic Umberto I of Rome. Written informed consent will be obtain from all eligible participants following complete description of study details. Participants will be informed regarding their freedom to withdraw from the trial anytime without any negative effect on their therapy. The trial will be registered at the Italian Registry of Clinical Trials.

Consecutively the investigators will enroll patients who met the diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5) with criteria of moderate to severe OCD and a Yale Brown Obsessive Compulsive Scale (Y-BOCS) score of >21 were selected to be in this study. Y-BOCS will be used to evaluate treatment efficacy. This is a well-validated 10-item rating scale, which is widely used to measure the severity of OCD symptoms. Participants were rated by Y-BOCS at baseline and at 2, 4, 6, 8, 10 and 12 months. During the screening period, T4 and T6 follow-up visits all participants will undergo an extensive neuropsychological evaluation. Speed processing by using the WAIS-IV Digit Symbol, attention by means of the Trial Making Test and a computerized alertness and Go/no go task memory by using the Digit and Corsi Span, a modified version of Corsi Block Tapping test, the Story recall of Rivermead Behavioral Memory Test and a modified version of Babcock Story recall test executive functions by means of Stroop Task, a modified version of Tower of London and the Modified Five Point Test.

Interventions:

This is a double blind, randomized, parallel group, placebo controlled, monocentric trial in subjects with OCD. The trial includes one active dose arm of Memantine and placebo.

The trial consists of four distinct periods:

* Screening: The screening period may last up to 4 weeks for each eligible patient.
* Thirty-two-week double-blind up-titration treatment period (from T0 to T4): After screening, patients who meet all eligibility criteria will be randomly assigned to one of two arms (Memantine or placebo) in a 1:1 ratio. Following baseline assessments, each patient will receive a daily administration of Memantine/placebo up to 20mg/day.
* Eight-week double-blind down-titration treatment period (from T4 to T5): At T4, the dose of Memantine/placebo will be reduced at 10mg/day due to safety reasons before the end of treatment (T5).
* Follow-up period (from T5 to T6): After the 40-week double-blind treatment period, patients will be asked to come back for the follow-up visit (T6) 8 weeks after the end of the treatment (T5).

Trial Design:

Placebo and memantine tablets will be identical in shapes, colors, weight and scent. In advance the investigators will prepared a random-number sequence that a computer-generated for random group assignment. Treatment allocation will be concealed from patients and physician will rated patients and from statistician. Separate individuals will be responsible for randomization and rating patients.

Sample size:

The investigators based the power calculation on previous study. Taking into account two groups and seven measurement time points, the minimum sample size will be 20 (calculated with G*Power 3.1).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis by a psychiatrist of current OCD according to the DSM 5
* patients in therapy with a stable SSRI for at least three weeks prior
* written informed consent.

Exclusion Criteria:

* Substance dependence
* IQ <70
* comorbid psychiatric disorders
* female pregnant or breast-feeding or intend to become pregnant during the period of the study
* concomitant treatments (rTMS, CBT, other glutamate-modulating drugs)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of OCD symptoms will be intended as a rate of more then 1/3 on the Y-BOCS total score. | From the week number 5 to the week number 52
  The investigators will evaluate the improvement of symptoms through a decrease of OCD, intended as a rate of more then 1/3 on the Y-BOCS total score.

SECONDARY OUTCOMES:
Evaluate the minimum effective dose of memantine | From the week number 5 to the week number 46
  The second aim of the study is to evaluate the minimum effective dose of memantine in these patients. The investigators will evaluate the improvement of symptoms through reduction of both subscales (obsessive thoughts and compulsive behaviors) and of the total Y-BOCS score.
Evaluate the effects after drug withdrawal through follow up | From the week number 5 to the week number 46
  Moreover the investigators will evaluate the effects after drug withdrawal during follow up through reduction of both subscales (obsessive thoughts and compulsive behaviors) and of the total Y-BOCS score.

OTHER OUTCOMES:
Improvement at the WAIS-IV. | from the week number 5 to the week number 52
  The third aim is to investigate the effect of memantine on patients without cognitive impairment, on improvement of cognitive functions through the reduction of total score of the WAIS-IV Digit Symbol.
Improvement at the Trial Making Test. | from the week number 5 to the week number 52
  The fourth aim is to evaluate the effect of memantine on patients without cognitive impairment, on improvement of cognitive functions through the reduction of total score of the Trial Making Test.
Improvement at the Digit and Corsi Span. | from the week number 5 to the week number 52
  The fifth aim is to evaluate the effect of memantine on patients without cognitive impairment, on improvement of cognitive functions through the reduction of total score of the Digit and Corsi Span.
Improvement at the Corsi Block Tapping test. | from the week number 5 to the week number 52
  The sixth aim is to evaluate the effect of memantine on patients without cognitive impairment, on improvement of cognitive functions through the reduction of total score of the Corsi Block Tapping test.
Improvement at the Story recall of Rivermead Behavioral Memory Test. | from the week number 5 to the week number 52
  The sixth aim is to evaluate the effect of memantine on patients without cognitive impairment, on improvement of cognitive functions through the reduction of total score of the Story recall of Rivermead Behavioral Memory Test.
Improvement at the Babcock Story recall test. | from the week number 5 to the week number 52
  The eighth aim is to evaluate the effect of memantine on patients without cognitive impairment, on improvement of cognitive functions through the reduction of total score of the Story recall of Babcock Story recall test.
Improvement at the Stroop Task. | from the week number 5 to the week number 52
  The ninth aim is to evaluate the effect of memantine on patients without cognitive impairment, on improvement of cognitive functions through the reduction of total score of the Stroop Task.
Improvement at the Tower of London. | from the week number 5 to the week number 52
  The tenth aim is to evaluate the effect of memantine on patients without cognitive impairment, on improvement of cognitive functions through the reduction of total score of the Tower of London.
Improvement at the the Modified Five Point Test. | from the week number 5 to the week number 52
  The eleventh aim is to evaluate the effect of memantine on patients without cognitive impairment, on improvement of cognitive functions through the reduction of total score of the the Modified Five Point Test.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruscio AM, Stein DJ, Chiu WT, Kessler RC. The epidemiology of obsessive-compulsive disorder in the National Comorbidity Survey Replication. Mol Psychiatry. 2010 Jan;15(1):53-63. doi: 10.1038/mp.2008.94. Epub 2008 Aug 26. PMID 18725912
- [Background] Stein DJ, Fineberg NA, Bienvenu OJ, Denys D, Lochner C, Nestadt G, Leckman JF, Rauch SL, Phillips KA. Should OCD be classified as an anxiety disorder in DSM-V? Depress Anxiety. 2010 Jun;27(6):495-506. doi: 10.1002/da.20699. PMID 20533366
- [Background] Phillips KA, Stein DJ, Rauch SL, Hollander E, Fallon BA, Barsky A, Fineberg N, Mataix-Cols D, Ferrao YA, Saxena S, Wilhelm S, Kelly MM, Clark LA, Pinto A, Bienvenu OJ, Farrow J, Leckman J. Should an obsessive-compulsive spectrum grouping of disorders be included in DSM-V? Depress Anxiety. 2010 Jun;27(6):528-55. doi: 10.1002/da.20705. PMID 20533367
- [Background] Burguiere E, Monteiro P, Mallet L, Feng G, Graybiel AM. Striatal circuits, habits, and implications for obsessive-compulsive disorder. Curr Opin Neurobiol. 2015 Feb;30:59-65. doi: 10.1016/j.conb.2014.08.008. Epub 2014 Sep 19. PMID 25241072
- [Background] Milad MR, Rauch SL. Obsessive-compulsive disorder: beyond segregated cortico-striatal pathways. Trends Cogn Sci. 2012 Jan;16(1):43-51. doi: 10.1016/j.tics.2011.11.003. Epub 2011 Dec 2. PMID 22138231
- [Background] Graybiel AM, Rauch SL. Toward a neurobiology of obsessive-compulsive disorder. Neuron. 2000 Nov;28(2):343-7. doi: 10.1016/s0896-6273(00)00113-6. No abstract available. PMID 11144344
- [Background] Ting JT, Feng G. Neurobiology of obsessive-compulsive disorder: insights into neural circuitry dysfunction through mouse genetics. Curr Opin Neurobiol. 2011 Dec;21(6):842-8. doi: 10.1016/j.conb.2011.04.010. Epub 2011 May 24. PMID 21605970
- [Background] Ninio J, Mizraji E. String analysis and energy minimization in the partition of DNA sequences. J Mol Biol. 1989 Jun 5;207(3):585-96. doi: 10.1016/0022-2836(89)90467-1. PMID 2760924
- [Background] Boedhoe PSW, Schmaal L, Abe Y, Alonso P, Ameis SH, Anticevic A, Arnold PD, Batistuzzo MC, Benedetti F, Beucke JC, Bollettini I, Bose A, Brem S, Calvo A, Calvo R, Cheng Y, Cho KIK, Ciullo V, Dallaspezia S, Denys D, Feusner JD, Fitzgerald KD, Fouche JP, Fridgeirsson EA, Gruner P, Hanna GL, Hibar DP, Hoexter MQ, Hu H, Huyser C, Jahanshad N, James A, Kathmann N, Kaufmann C, Koch K, Kwon JS, Lazaro L, Lochner C, Marsh R, Martinez-Zalacain I, Mataix-Cols D, Menchon JM, Minuzzi L, Morer A, Nakamae T, Nakao T, Narayanaswamy JC, Nishida S, Nurmi E, O'Neill J, Piacentini J, Piras F, Piras F, Reddy YCJ, Reess TJ, Sakai Y, Sato JR, Simpson HB, Soreni N, Soriano-Mas C, Spalletta G, Stevens MC, Szeszko PR, Tolin DF, van Wingen GA, Venkatasubramanian G, Walitza S, Wang Z, Yun JY; ENIGMA-OCD Working Group; Thompson PM, Stein DJ, van den Heuvel OA; ENIGMA OCD Working Group. Cortical Abnormalities Associated With Pediatric and Adult Obsessive-Compulsive Disorder: Findings From the ENIGMA Obsessive-Compulsive Disorder Working Group. Am J Psychiatry. 2018 May 1;175(5):453-462. doi: 10.1176/appi.ajp.2017.17050485. Epub 2017 Dec 15. PMID 29377733
- [Background] Marinova Z, Chuang DM, Fineberg N. Glutamate-Modulating Drugs as a Potential Therapeutic Strategy in Obsessive-Compulsive Disorder. Curr Neuropharmacol. 2017;15(7):977-995. doi: 10.2174/1570159X15666170320104237. PMID 28322166
- [Background] Lovinger DM. Neurotransmitter roles in synaptic modulation, plasticity and learning in the dorsal striatum. Neuropharmacology. 2010 Jun;58(7):951-61. doi: 10.1016/j.neuropharm.2010.01.008. Epub 2010 Jan 21. PMID 20096294
- [Background] Gillan CM, Papmeyer M, Morein-Zamir S, Sahakian BJ, Fineberg NA, Robbins TW, de Wit S. Disruption in the balance between goal-directed behavior and habit learning in obsessive-compulsive disorder. Am J Psychiatry. 2011 Jul;168(7):718-26. doi: 10.1176/appi.ajp.2011.10071062. Epub 2011 May 15. PMID 21572165
- [Background] Chakrabarty K, Bhattacharyya S, Christopher R, Khanna S. Glutamatergic dysfunction in OCD. Neuropsychopharmacology. 2005 Sep;30(9):1735-40. doi: 10.1038/sj.npp.1300733. PMID 15841109
- [Background] Bhattacharyya S, Khanna S, Chakrabarty K, Mahadevan A, Christopher R, Shankar SK. Anti-brain autoantibodies and altered excitatory neurotransmitters in obsessive-compulsive disorder. Neuropsychopharmacology. 2009 Nov;34(12):2489-96. doi: 10.1038/npp.2009.77. Epub 2009 Aug 12. PMID 19675532
- [Background] Arnold PD, Rosenberg DR, Mundo E, Tharmalingam S, Kennedy JL, Richter MA. Association of a glutamate (NMDA) subunit receptor gene (GRIN2B) with obsessive-compulsive disorder: a preliminary study. Psychopharmacology (Berl). 2004 Aug;174(4):530-8. doi: 10.1007/s00213-004-1847-1. Epub 2004 Apr 9. PMID 15083261
- [Background] Shin DJ, Jung WH, He Y, Wang J, Shim G, Byun MS, Jang JH, Kim SN, Lee TY, Park HY, Kwon JS. The effects of pharmacological treatment on functional brain connectome in obsessive-compulsive disorder. Biol Psychiatry. 2014 Apr 15;75(8):606-14. doi: 10.1016/j.biopsych.2013.09.002. Epub 2013 Oct 4. PMID 24099506
- [Background] Niciu MJ, Henter ID, Luckenbaugh DA, Zarate CA Jr, Charney DS. Glutamate receptor antagonists as fast-acting therapeutic alternatives for the treatment of depression: ketamine and other compounds. Annu Rev Pharmacol Toxicol. 2014;54:119-39. doi: 10.1146/annurev-pharmtox-011613-135950. PMID 24392693
- [Background] Murphy DL, Moya PR, Fox MA, Rubenstein LM, Wendland JR, Timpano KR. Anxiety and affective disorder comorbidity related to serotonin and other neurotransmitter systems: obsessive-compulsive disorder as an example of overlapping clinical and genetic heterogeneity. Philos Trans R Soc Lond B Biol Sci. 2013 Feb 25;368(1615):20120435. doi: 10.1098/rstb.2012.0435. Print 2013. PMID 23440468
- [Background] Andrade C. Augmentation With Memantine in Obsessive-Compulsive Disorder. J Clin Psychiatry. 2019 Dec 3;80(6):19f13163. doi: 10.4088/JCP.19f13163. PMID 31846244
- [Result] Pittenger C, Krystal JH, Coric V. Glutamate-modulating drugs as novel pharmacotherapeutic agents in the treatment of obsessive-compulsive disorder. NeuroRx. 2006 Jan;3(1):69-81. doi: 10.1016/j.nurx.2005.12.006. PMID 16490414
- [Result] Parsons CG, Danysz W, Quack G. Memantine is a clinically well tolerated N-methyl-D-aspartate (NMDA) receptor antagonist--a review of preclinical data. Neuropharmacology. 1999 Jun;38(6):735-67. doi: 10.1016/s0028-3908(99)00019-2. PMID 10465680
- [Result] Haghighi M, Jahangard L, Mohammad-Beigi H, Bajoghli H, Hafezian H, Rahimi A, Afshar H, Holsboer-Trachsler E, Brand S. In a double-blind, randomized and placebo-controlled trial, adjuvant memantine improved symptoms in inpatients suffering from refractory obsessive-compulsive disorders (OCD). Psychopharmacology (Berl). 2013 Aug;228(4):633-40. doi: 10.1007/s00213-013-3067-z. Epub 2013 Mar 23. PMID 23525525
- [Result] Ghaleiha A, Entezari N, Modabbernia A, Najand B, Askari N, Tabrizi M, Ashrafi M, Hajiaghaee R, Akhondzadeh S. Memantine add-on in moderate to severe obsessive-compulsive disorder: randomized double-blind placebo-controlled study. J Psychiatr Res. 2013 Feb;47(2):175-80. doi: 10.1016/j.jpsychires.2012.09.015. Epub 2012 Oct 9. PMID 23063327
- [Result] Modarresi A, Sayyah M, Razooghi S, Eslami K, Javadi M, Kouti L. Memantine Augmentation Improves Symptoms in Serotonin Reuptake Inhibitor-Refractory Obsessive-Compulsive Disorder: A Randomized Controlled Trial. Pharmacopsychiatry. 2018 Nov;51(6):263-269. doi: 10.1055/s-0043-120268. Epub 2017 Nov 3. PMID 29100251
- [Derived] Maraone A, Trebbastoni A, Di Vita A, D'Antonio F, De Lena C, Pasquini M. Memantine for Refractory Obsessive-Compulsive Disorder: Protocol for a Pragmatic, Double-blind, Randomized, Parallel-Group, Placebo-Controlled, Monocenter Trial. JMIR Res Protoc. 2023 May 11;12:e39223. doi: 10.2196/39223. PMID 37166948